CLINICAL TRIAL: NCT03555045
Title: The Effect of Slanted Recession of Horizontal Muscle on Horizontal Strabismus With Abnormal Accommodative Convergence /Accommodation Ratio (AC/A)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96302
Record Dates: First submitted 2018-04-11; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-01

CONDITIONS: Horizontal Strabismus With High AC/A Ratio

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conducting the slanted recession technique (Active Comparator): conducting the slanted recession technique on the superior and inferior poles of the muscle based on far and near deviations.
  Interventions: Procedure: conducting the slanted recession technique on the superior and inferior poles
- conducting the augmented recession technique on the muscle (Active Comparator): conducting the augmented recession technique on the muscle for 1 to 1.50 mm more compared with the standard method.
  Interventions: Procedure: conducting the augmented recession technique on the muscle

INTERVENTIONS:
Procedure: conducting the slanted recession technique on the superior and inferior poles — conducting the slanted recession technique on the superior and inferior poles of the muscle based on far and near deviations.
  Arms: conducting the slanted recession technique
Procedure: conducting the augmented recession technique on the muscle — conducting the augmented recession technique on the muscle for 1 to 1.50 mm more compared with the standard method.
  Arms: conducting the augmented recession technique on the muscle

SUMMARY:
Different methods was tried to treat high AC/A strabismus cases;such as prescription of bifocal glasses in esotropia,recession of horizontal muscles with posterior fixation sutures,more recession than needed for far deviation(augmented recession),recession and pulley fixation and slant recession.

Different results was reported for any type of above methods. In recent studies,slanted recession was applied for high AC/A in esotropic cases and success rate of 67% was reported.but there was no unanimity for procedure of choice.

Since slant recession method is simpler and has low side effect than the other methods,therefore in this study the investigators want to peruse the outcome of this method on high AC/A horizontal strabismus.

ELIGIBILITY:
Inclusion Criteria:

* all patients with horizontal strabismus that the different between far deviation and near deviation is more than 10 pd

Exclusion Criteria:

* all patients who had history of surgery on horizontal muscles and patients with pseudo high AC/A ratio.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
far-near deviation difference | 90 days after surgery
  difference between the far and near deviations

SECONDARY OUTCOMES:
success rate of surgery | 90 days after surgery
  in cases with difference of far and near deviation less than 10 prism diopters

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran